CLINICAL TRIAL: NCT02461667
Title: Comparative Evaluation of Subgingivally Delivered 1% Metformin and 1% Alendronate Gel in Treatment of Chronic Periodontitis: a Randomized Placebo Controlled Clinical Trial
Brief Title: Alendronate Compared to Metformin in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and head, Dept. of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014G
Record Dates: First submitted 2015-05-19; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Periodontitis
Keywords: alendronate, metformin
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): SRP plus placebo SRP was done for all the subjects. Placebo gel was delivered subgingivally into the pocket
  Interventions: Drug: SRP plus Placebo Gel
- Metformin (Active Comparator): SRP plus Metformin SRP was done for all the subjects. metformin was delivered in the pocket subgingivally
  Interventions: Drug: SRP plus Metformin gel
- Alendronate (Active Comparator): SRP plus Alendronate SRP was done for all the subjects. Alendronate was delivered in the pocket subgingivally
  Interventions: Drug: SRP plus Alendronate gel

INTERVENTIONS:
Drug: SRP plus Placebo Gel — After SRP, placebo gel was delivered subgingivally into the pocket
  Other Names: Placebo
  Arms: placebo
Drug: SRP plus Alendronate gel — Alendronate (ALN) After SRP, ALN gel was delivered subgingivally into the pocket
  Other Names: Alendronate gel
  Arms: Alendronate
Drug: SRP plus Metformin gel — Metformin (MF) After SRP, MF gel was delivered subgingivally into the pocket
  Other Names: Metformin gel
  Arms: Metformin

SUMMARY:
This is a 9 month randomised controlled clinical comparing the clinical efficacy of 1%metformin and 1%alendronate in chronic periodontitis subjects.

DETAILED DESCRIPTION:
ABSTRACT Background: Since Metformin (MF) induces osteoblast growth and differentiation while Alendronate (ALN) act as an antiosteolytic agent. The aim of the present study is to evaluate and compare the efficacy of 1% ALN and 1% MF gel as a local drug delivery system in adjunct to scaling and root planing (SRP) for the treatment of intrabony defects in patients with chronic periodontitis.

Methods:

The study had 3 groups comprising of ninety subjects, divided into three groups 1% MF with SRP, 1% ALN with SRP and placebo gel with SRP. Clinical parameters (plaque index (PI), modified sulcus bleeding index (mSBI), probing pocket depth (PPD), and clinical attachment level (CAL) were recorded at baseline, 3, 6 and 9 months. Radiographic parameters intrabony defect depth (IBD) and defect depth reduction (DDR%) was calculated on standardized radiographs by using image analysis software at 6 and 9 months

ELIGIBILITY:
Inclusion Criteria:

* All the subjects were systemically healthy
* subjects with sites having CAL ≥ 3 mm, PPD ≥ 5 mm,
* vertical bone loss ≥ 3 mm on intraoral periapical radiographs (IOPA) and
* subjects with no history of periodontal intervention in the last 6 months.

Exclusion Criteria:

* patients with systemic diseases like cardiovascular disease
* diabetes or HIV infection or on medications like corticosteroids which may impede the healing in periodontal tissues.
* pregnant/lactating females
* tobacco users
* alcoholics
* patients with unsatisfactory oral hygiene (plaque index greater than 1.5)
* teeth having gingival recession, caries involving pulp, intrabony defect present interproximally, grade 2/3 mobility
* Furthermore, patients allergic to Metformin and alendronate or those taking Metformin and alendronate systemically were excluded.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
bone fill | baseline to 9 months
  amount of bone fill from baseline to 9 months

SECONDARY OUTCOMES:
Relative vertical clinical attachment level | baseline to 9 months
  change in Relative vertical clinical attachment level baseline to 9 months
probing depth | baseline to 9 months
  change in probing depth from baseline to 9 months